CLINICAL TRIAL: NCT03912740
Title: Effect of Dexmedetomidine vs 0.9% Sodium Chloride on Nol-Index Guided Remifentanil Analgesia: a Double-blinded Bicenter Randomized Controlled Trial
Brief Title: Effect of Dexmedetomidine on Nol-Index Guided Remifentanil Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Collaborators: Saint-Pierre University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P2018/568
Record Dates: First submitted 2019-02-25; First posted 2019-04-11 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Nociceptive Pain; Anesthesia; Opioid Use; Perioperative/Postoperative Complications
MeSH Terms: conditions — Nociceptive Pain; Postoperative Complications | interventions — Dexmedetomidine; Sodium Chloride; Saline Solution; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remifentanil Analgesia (Active Comparator): Continuous intraoperative analgesia with remifenanil + 0.9% sodium chloride
  Interventions: Drug: sodium chloride; Drug: Remifentanil
- Remifentanil and Dexmedetomidine Analgesia (Active Comparator): Continuous intraoperative analgesia with remifenanil + dexmedetomidine
  Interventions: Drug: Dexmedetomidine; Drug: Remifentanil

INTERVENTIONS:
Drug: Dexmedetomidine — Patients in the dexmedetomidine-remifentanil group will receive an infusion of 0.6 mcg/kg in half an hour followed by an infusion of 0.6 mcg/kg/hour.
  Other Names: Dexdor
  Arms: Remifentanil and Dexmedetomidine Analgesia
Drug: sodium chloride — Patients in the remifentanil group will receive an infusion of 0.9% sodium chloride instead of dexmedetomidine (identical infusion rate)
  Other Names: normal saline 0.9%
  Arms: Remifentanil Analgesia
Drug: Remifentanil — Both groups will have remifentanil analgesia guided by the Nol-Index
  Other Names: Ultiva

SUMMARY:
Background:

Analgesia remains to this day a challenge for anesthesiologists. Dexmedetomidine, a potent central alpha-2 agonist, has been shown to have analgesic and opioid sparing effects. The classic analgesic strategy focuses on opioid administration guided by estimated time of elimination and hemodynamic response (increase in blood pressure and heart rate). This technique is not sensitive and forces the anesthesiologist to be one step behind nociception, the patient's unconscious response to pain.

PMD-200 (Medasense, Israel) displays the Nociceptive level (NOL)-Index as marker of nociception. The NOL-Index ranges from 0 (no nociception) to 100 (intense nociception) and the recommended analgesic range during surgery is from 10 to 25 (Medasense recommendations).

The goal of this study is to compare two analgesia strategies guided by the NOL Index (range 10-25) using either remifentanil TCI (target controlled infusion) alone or remifentanil TCI associated with a continuous dexmedetomidine infusion.

Methods:

A total of 100 patients will be included and informed consent will be acquired. This bi-center study will take place at Erasme University Hospital (primary center) and Saint-Pierre University Hospital. Patients will be randomized into either two groups: remifentanil and placebo versus remifentanil and dexmedetomidine. Both groups will be monitored using the PMD-200 that will guide the analgesic therapy strategy. Investigators and patients will be blinded to dexmedetomidine and placebo administration. The primary outcome will be intraoperative remifentanil consumption. Secondary outcomes will include postoperative opioid administration, opioid associated complications, hemodynamics, and hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

- American Society of Anesthesiologists (ASA) grades 1-2 undergoing scheduled stomatological, cervical, and thyroid surgery anticipated to last at least two hours

Exclusion Criteria:

* ASA score >2
* Preoperative organ dysfunction
* Patients with non-regular cardiac rhythm
* Implanted pacemakers
* Emergent surgery
* Pregnancy or lactation
* Allergy or intolerance to any of the study drugs
* Participation in another interventional study
* Patient refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Remifentanil consumption measured as the amount (µg) of remifentanil administered during the anesthestic | 6 hours
  Intraoperative remifentanil consumption

SECONDARY OUTCOMES:
Propofol Consumption measured as the amount of propofol (mg) administered during the anesthestic | 6 hours
  Intraoperative propofol consumption
Use of vasoactive drugs | 6 hours
  Use and amount of vasoactive drugs used (ephedrine/phenylephrine/noradrenaline)
Use of hypotensive drugs | 6 hours
  Use and amount of hypotensive drugs used (nicardipine/esmolol)
Net fluid balance | 6 hours
  Sum of in (infused fluids) and out (net blood loss, diuresis, other losses)
Time to extubation | 6 hours
  Time from end of surgery to extubation of patient
Number of patients with intraoperative hypotension | 6 hours
  Intraoperative MAP (mean arterial pressure) <65 mmHg*
  * Patients that have chronic hypertension or that are 65 years of age or older will have a MAP threshold of 75mmHg (and not 65mmHg).
Number of patients with intraoperative hypertension | 6 hours
  Intraoperative MAP≥100 or surgical need to decrease blood pressure
Number of patients with hemodynamic instability | 6 hours
  MAP<65 mmHg*, HR<45, MAP≥100, HR>90
  * Patients that have chronic hypertension or that are 65 years of age or older will have a MAP threshold of 75mmHg for hypotension (and not 65mmHg).
Intraoperative heart rate | 6 hours
  Measurement during key intraoperative periods (before induction, after induction, after intubation, before incision, after incision, every 15 minutes after incision, after end of surgery, and after reversal of anesthesia)
Intraoperative blood pressure | 6 hours
  Measurement during key intraoperative periods (before induction, after induction, after intubation, before incision, after incision, every 15 minutes after incision, after end of surgery, and after reversal of anesthesia)
Intraoperative Nol-Index | 6 hours
  Measurement during key intraoperative periods (before induction, after induction, after intubation, before incision, after incision, every 15 minutes after incision, after end of surgery, and after reversal of anesthesia)
Intraoperative remifentanil target cite concentration | 6 hours
  Measurement during key intraoperative periods (before induction, after induction, after intubation, before incision, after incision, every 15 minutes after incision, after end of surgery, and after reversal of anesthesia)
Postoperative morphine consumption | 24 hours
  mg of morphine administered postoperatively
Number of patients with postoperative opioid-related side effect (composite and individual complications) | 72 hours
  Post-operative nausea or vomiting within the first 24 h, postoperative hypoxemia (need within 24h postop to have supplemental oxygen (to maintain sat >94%), and pruritus.
PACU length of stay (LOS) | 48 hours
  hours spent at PACU
Hospital LOS | 28 days
  days spents hospitalized

CONTACTS AND LOCATIONS:
Overall Officials: Sean Coeckelenbergh, M.D., Principal Investigator — Université Libre de Bruxelles
Locations (1):
- Erasme University Hospital, Brussels, Belgium

REFERENCES:
- [Derived] Coeckelenbergh S, Doria S, Patricio D, Perrin L, Engelman E, Rodriguez A, Di Marco L, Van Obbergh L, Estebe JP, Barvais L, Kapessidou P. Effect of dexmedetomidine on Nociception Level Index-guided remifentanil antinociception: A randomised controlled trial. Eur J Anaesthesiol. 2021 May 1;38(5):524-533. doi: 10.1097/EJA.0000000000001402. PMID 33259449